CLINICAL TRIAL: NCT03992261
Title: Open Label Evaluation of the Adrenal Suppression Potential and Pharmacokinetic Properties of Twice Daily Halobetasol Propionate Foam, 0.05% in Subjects 12 to Less Than 18 Years of Age With Plaque Psoriasis Receiving Two Weeks of Treatment
Brief Title: Adrenal Suppression and Absorption Study of Halobetasol Propionate Foam in Subjects 12-17 With Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayne Pharma International Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 122-0551-209
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-03

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Halobetasol Propionate Foam (Experimental): 2 weeks of application, 2 times daily
  Interventions: Drug: Halobetasol Topical Foam

INTERVENTIONS:
Drug: Halobetasol Topical Foam — Foam
  Other Names: HBP Foam

SUMMARY:
The purpose of this study is to evaluate Halobetasol Propionate (HBP) foam, 0.05% in subjects aged 12 through less than 18 years with plaque psoriasis in order to check the safety, the potential to suppress the adrenal glands and the degree to which the drug is absorbed into the bloodstream.

DETAILED DESCRIPTION:
This is a Phase 4 (for US site only, Phase 2 for non-US sites), open label, multicenter study of halobetasol propionate (HBP) Foam, 0.05% in male and female subjects who are 12 to less than 18 years of age with stable plaque psoriasis. Twenty-four subjects with stable plaque psoriasis on at least 10% of their body surface area (BSA) (excluding the face, scalp, groin, axillae, and other intertriginous areas), who fulfill the inclusion/exclusion criteria will be enrolled at multiple study sites in the US and Europe. All subjects are to have a Cosyntropin Stimulation Test (CST) to assess their (hypothalmic pituitary adrenal) HPA axis response at Visit 1/Screening initiated between 7 and 9 AM. Enrollment into the treatment phase of the study will be timed such that the Screening CST is performed a minimum of 20 days before Visit 2/Baseline. At Visit 2/Baseline, eligible subjects with normal adrenal function will be eligible to participate in the study.

The primary objective of the study is to assess safety, not efficacy. Safety will be determined by assessing the adrenal suppression potential and the PK properties of HBP Foam, 0.05% applied twice daily in male and female subjects who were 12 to less than 18 years of age with stable plaque psoriasis.

Other safety endpoints include plasma levels of HBP. Trough HBP concentrations in plasma on day 8 and 15 will be calculated and summarized. Efficacy will also be noted utilizing the Investigator's Global Assessment (IGA) scale and percent BSA treated and affected with disease to assess and document any changes observed with regard to IGA and percent BSA.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject is male or non-pregnant female and is 12 to less than 18 years of age
* Subject has provided written informed assent and was accompanied by the parent or legal guardian at the time of assent/consent signing
* Subject has a clinical diagnosis of stable plaque psoriasis involving a minimum of 10% Body Surface Area (BSA)
* Subject has an Investigator's Global Assessment (IGA) score of at least three (3 = moderate) at the Baseline Visit

Key Exclusion Criteria:

* Subject has spontaneously improving or rapidly deteriorating plaque psoriasis
* Subject has guttate, pustular, erythrodermic or other non-plaque forms of psoriasis
* Subject has a physical condition which, in the investigator's opinion, might impair evaluation of plaque psoriasis, adrenal axis function or which exposes the subject to an unacceptable risk by study participation
* Subject has had prolonged exposure to natural or artificial sources of ultraviolet radiation
* Subject is pregnant, lactating, or is planning to become pregnant during the study
* Subject is currently enrolled in an investigational drug or device study

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Piacquadio, MD, Study Director — Therapeutics, Inc.
Locations (11):
- United States (2):
  - Investigative Site 2, Hialeah, Florida
  - Investigative Site 1, Saint Joseph, Missouri
- Georgia (3):
  - Investigative Site 9, Batumi
  - Investigative Site 10, Tbilisi
  - Investigative Site 11, Tbilisi
- Poland (3):
  - Investigative Site 3, Krakow
  - Investigative Site 5, Tarnów
  - Investigative Site 4, Warsaw
- Ukraine (3):
  - Investigative Site 8, Rivne
  - Investigative Site 6, Uzhhorod
  - Investigative Site 7, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Groups:
- Halobetasol Propionate Foam, 0.05%: 24 subjects with stable plaque psoriasis on at least 10% body surface area (BSA) (excluding: face, scalp, groin, axillae, and other intertriginous areas), who fulfilled the inclusion/exclusion criteria were enrolled at multiple study sites in the US and Europe. All subjects were to have a Cosyntropin Stimulation Test (CST) to assess their hypothalamic pituitary adrenal (HPA) axis response at Visit 1/Screening initiated between 7 and 9 AM. Enrollment into the treatment phase of the study should have been timed such that the Screening CST was performed a minimum of 20 days before Visit 2/Baseline. At Visit 2/Baseline, eligible subjects with normal adrenal function were eligible to participate in the study.
  Subjects were instructed to apply Halobetasol Propionate (HBP) Foam, 0.05% to all psoriasis plaques identified at Visit 2/Baseline twice daily (approximately every 12 hours) for the assigned treatment period or until the investigator verified the subject's psoriasis had cleared.
Period: Overall Study
Arm/Group | Halobetasol Propionate Foam, 0.05%
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Halobetasol Propionate Foam: Open label evaluation all participants received Halobetasol Propionate Foam, 0.05% 2 times daily for 2 weeks of application in subjects 12-17 years of age
Arm/Group | Halobetasol Propionate Foam
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects to Exhibit Adrenal Suppression as Measured by a Cosyntropin Stimulation Test
Description: A subject is considered to have adrenal suppression evidence if post cosyntropin stimulation lab draw result is less than or equal to 18.0 mcg/100 mL.
  HPA axis responses to cosyntropin were dichotomized to normal and abnormal. Cosyntropin stimulation testing was performed at Screening and Day 15 and approximately 4 weeks post-treatment if a subject's laboratory results at Day 15 showed an abnormal hypothalamic pituitary adrenal (HPA) axis response (HPA axis suppression). An abnormal HPA axis response was defined as a 30-minute post-stimulation serum cortisol level of ≤18 μg/dL at end of study (EOS).
Time Frame: Screening, Day 15, and approximately 4 weeks post-treatment, an average of 28 days
Population: Evaluable subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Halobetasol Propionate Foam
Number analyzed (Participants) | 23
Participants
  Abnormal HPA Axis Response | 6
  Normal HPA Axis Response | 17

2. Primary Outcome: Plasma Concentration of HBP at Screening, Day 8 and Day 15
Description: Morning trough concentrations of HBP in plasma at Screening, Day 8, and Day 15 were summarized for the PK population using geometric mean, coefficient of variation in addition to n, mean, median, standard deviation (SD), minimum, and maximum.
Time Frame: 15 days
Population: Pharmacokinetic Population
Measure: Count of Participants; unit: Participants
Groups:
- Halobetasol Propionate Foam, 0.05%: 24 subjects with stable plaque psoriasis on at least 10% BSA (excluding: face, scalp, groin, axillae, and other intertriginous areas), who fulfilled the inclusion/exclusion criteria were enrolled at multiple study sites in the US and Europe. All subjects were to have a Cosyntropin Stimulation Test (CST) to assess their HPA axis response at Visit 1/Screening initiated between 7 and 9 AM. Enrollment into the treatment phase of the study should have been timed such that the Screening CST was performed a minimum of 20 days before Visit 2/Baseline. At Visit 2/Baseline, eligible subjects with normal adrenal function were eligible to participate in the study.
  Subjects were instructed to apply HBP Foam, 0.05% to all psoriasis plaques identified at Visit 2/Baseline twice daily (approximately every 12 hours) for the assigned treatment period or until the investigator verified the subject's psoriasis had cleared.
Arm/Group | Halobetasol Propionate Foam, 0.05%
Number analyzed (Participants) | 23
Participants
  Baseline number of participants with plasma morning trough concentrations below limits | 23
  Day 8 number of participants with plasma morning trough concentrations below limits | 14
  Day 15/EOS number of participants with plasma morning trough concentrations below limits | 13
  Day 8 Subjects with measurable levels of HBP at morning trough | 9
  Day 15/EOS Subjects with measurable levels of HBP at morning trough | 6
Statistical Analysis 1: Comparison: Halobetasol Propionate Foam, 0.05%; Outcome measure: extent of exposure, HPA axis suppression, and pharmacokinetic analysis; Test type: Other — Mean, median, SD, minimum/maximum determined for total amount of test article used by each subject in Safety, Evaluable, and PK populations HPA Axis Suppression: Proportion of subjects manifesting laboratory evidence of adrenal suppression at EOS were presented with 95% confidence intervals (CIs) for Evaluable and Safety populations. Descriptive statistics for daily dose of test article were tabulated separately for suppressed and non-suppressed subjects. PK: Screening, Day 8, Day 15; p = 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Collected at study visits, days 1, 8, and 15.
Description: In accordance with standard MedDRA reporting requirements.
Arm/Group | Halobetasol Propionate Foam, 0.05%
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 7/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Halobetasol Propionate Foam, 0.05% (N=24)
Local skin reactions (Skin and subcutaneous tissue disorders) | 6 (6) — Telangiectasia and skin atrophy
ACTH Stimulation Test Abnormal (Endocrine disorders) | 7 (8) — ACTH Stimulation Test Abnormal

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT03992261/Prot_SAP_000.pdf